CLINICAL TRIAL: NCT03350568
Title: Study 1: Dietary Non Enzymatic Antioxidant Capacity and the Risk of Myocardial Infarction - The Swedish National March Cohort; Study 2: Dietary Total Antioxidant Capacity and Risk of Osteoarthritis in the Swedish National March Cohort
Brief Title: Dietary Antioxidants and Chronic Diseases-The Swedish National March Cohort
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ylva Trolle Lagerros, MD, Associate Professor, Karolinska Institutet
Other Study IDs: 97-205
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Myocardial Infarction; Diet; Osteoarthritis
Keywords: Antioxidants; Oxidative Stress; Atherosclerosis; Epidemiology
MeSH Terms: conditions — Myocardial Infarction; Osteoarthritis; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Total dietary NEAC assessed at baseline

SUMMARY:
Dietary antioxidants might protect from the development of chronic diseases by reducing levels of oxidative stress. The investigators therefore investigated the effect of dietary Non Enzymatic Antioxidant Capacity, which measures interactions between antioxidants in the whole diet, on the risk of 1) myocardial infarction and 2) osteoarthritis.

DETAILED DESCRIPTION:
Aim: Among an initial sample of 43,880 men and women who participated in the Swedish National March Cohort in 1997 the investigators aimed to investigate the effect of dietary Non Enzymatic Antioxidant Capacity (NEAC), assessed by a validated food frequency questionnaire at baseline, on the risk of 1) myocardial infarction and 2) osteoarthritis.

Identification of cases: Incident cases of myocardial infarction (ICD-10 code I21) and osteoarthritis (ICD-10 M15-19) were identified through exact linkages to the Swedish registries of population, migration, death, cancer, and inpatient care, using the national registration numbers as identifiers.

Main methods: The investigators fitted Cox proportional hazards regression models with age as underlying time scale to estimate hazard ratios (HR) with 95% confidence intervals (95% CI) for each outcome of interest at different levels of dietary NEAC. The investigators fitted multiple imputation models based on chained equations to address missingness of confounder variables.

ELIGIBILITY:
Exclusion Criteria Study 1:

* Incorrect national registration number
* Subjects who were <18 years
* Emigration before beginning of follow-up
* Death before beginning of follow-up
* Cancer diagnosis
* Any cardiovascular disease
* Extreme energy intake

Exclusion Criteria Study 2:

* Incorrect national registration number
* Subjects who were <40 years
* Emigration before beginning of follow-up
* Death before beginning of follow-up
* Osteoarthritis diagnosis
* Bone cancer- or metastases
* Joint injury or any arthropathy disease other than osteoarthritis
* Extreme energy intake

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study 1: Study population (n=34,543) was between the age of 18-94 years and free from cancer (except non-melanoma skin cancer) or any cardiovascular disease before the beginning of follow up.
  Study 2: Study population (n=29,188) was between the age of 40-94 years and free from osteoarthritis, bone cancer or -metastases , joint injury, or any arthropathy disease other than.
Sampling Method: Non-Probability Sample
Enrollment: 43880 (Actual)
Dates: Start 1997-10-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Myocardial Infarction | October 1, 1997-December 31, 2010
  Based on ICD-10 I21
Osteoarthritis | October 1, 1997-December 31, 2010
  Based on ICD-10 M15-19

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Trolle Lagerros, MD, PhD, Principal Investigator — Department of Medicine, Clinical Epidemiology, Karolinska Institutet; Department of Medicine, Clinic of Endocrinology, Karolinska University Hospital
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No